CLINICAL TRIAL: NCT03053908
Title: Orexin and Tau Pathology in Cognitively Normal Elderly (A New Prevention Strategy for Alzheimer's Disease)
Brief Title: Orexin and Tau Pathology in Cognitively Normal Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01529
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Elderly; Alzheimer Disease
Keywords: Orexin; Core Body Temperature
MeSH Terms: conditions — Alzheimer Disease | interventions — Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elderly Patients (Experimental)
  Interventions: Procedure: Actigraphy; Procedure: Nocturnal Polysomnograpahy (NPSG)

INTERVENTIONS:
Procedure: Actigraphy — Recording of sleep/wake cycle and TST by actigraphy to be completed at home by subject over 7 days
Procedure: Nocturnal Polysomnograpahy (NPSG) — N1 habituation and N2 data collection

SUMMARY:
Alzheimer's disease (AD) is a common neurodegenerative disease characterized by the accumulation of amyloid plaques and neurofibrillary tangles. Current consensus is that the AD pathological process begins decades before clinical symptoms occur. This long "preclinical" phase of AD might first become detectable in middle-age as deposits of hyperphosphorylated tau (P-tau) in the transentorhinal cortex and subcortical nuclei such as the locus coeruleus (LC) and the nucleus basalis of Meynert. There is strong preliminary evidence showing that cerebrospinal fluid (CSF) levels of orexin-A (OxA) are associated with increased P-tau (r=.52, p<.01) and total-tau (T-tau) (r=.42, p<.01) in cognitively normal older adults (mean age: 69.6±8.6 years).

This study poses that onset of tauopathy in the LC results in down regulation of orexin receptors, leading to a homeostatic increase of OxA production by the hypothalamus, which results in changes in core body temperature (CBT) and sleep disruption that cause further neurodegeneration. This hypothesis will be tested by demonstrating that increases in CSF P-tau are associated in vivo with tau PET uptake, and that tau binding in the LC is associated with increases in CSF OxA (Aim 1); and second, by analyzing the downstream consequences of increased central nervous system (CNS) OxA on sleep architecture and CBT (Aim 2). To test these hypotheses, 19 older adults (age 55-75) balanced by sex, will first perform a full clinical evaluation and PET-MRI where Tau burden will be analyzed by PET-MR using 18F-MK6240 (visits 1-2). Subjects will later undergo 7 days of actigraphy followed by nocturnal polysomnography (NPSG) for 2 consecutive nights (N1-2) during which we will measure CBT (visits 3-4). A morning lumbar puncture (LP) will be performed after N2 to obtain CSF.

DETAILED DESCRIPTION:
There is the potential to identify: 1) an association between CSF P-tau and in vivo 18F-MK6240 uptake; 2) a mechanism by which tau pathology may contribute to orexin dysfunction; 3) evidence that orexin dysfunction disrupts sleep and CBT rhythm; and, 4) CNS orexin dysfunction as a new therapeutic target for AD prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with normal cognition and 55-75 years of age will be enrolled.
* Subjects will be within normal limits on neurological and psychiatric examinations. All subjects enrolled will have both a Clinical Dementia Rating (CDR)=0 and a MMSE≥27
* All subjects will have had a minimum of 12 years of education. Among minority subjects >80% of the elderly individuals coming to the NYU-ADC meet this criterion. (The education restriction reduces performance variance on cognitive test measures and improves the sensitivity for detecting pathology and disease progression using the robust norms available at NYU. Given the majority of subjects will meet this criterion we do not consider this a major selection bias or generalization limitation for this study).
* An informed family member or life-partner (preferably bed-partner) will be interviewed over the phone or on the first or second visit to confirm the reliability of the subject interview.

Exclusion Criteria:

* History of brain tumor, MRI evidence of brain damage or brain disease including significant trauma, hydrocephalus, seizures, mental retardation or other serious neurological disorder (e.g. Parkinson's disease or other movement disorders). Subjects with a Fazekas scale >2 will be excluded109.
* Significant history of alcoholism or drug abuse.
* History of psychiatric illness (e.g., schizophrenia, bipolar, PTSD, or life-long history of major depression).
* Geriatric Depression Scale (short form)>5.
* Insulin dependent diabetes.
* Evidence of clinically relevant cardiac, pulmonary, endocrine or hematological conditions (e.g. low platelet levels).
* Physical impairment of such severity as to adversely affect the validity of psychological testing.
* Any prosthetic devices (e.g., pacemaker or surgical clips) that constitutes a hazard for MRI imaging or CBT measurements.
* History of a first-degree family member with early onset (age <60 years) dementia.
* Irregular sleep-wake rhythms (based on the actigraphy recordings) or significant OSA (AHI4%≥15).
* Medications affecting cognition or sleep.
* Presence of any known or suspected obstructive disease of the gastrointestinal tract, including but not limited to diverticulitis and inflammatory bowel disease.
* History of disorders or impairment of the gag reflex.
* Previous gastrointestinal surgery.
* Previous felinization of the esophagus.
* Subjects who might undergo Nuclear Magnetic Resonance (NMR) or MRI scanning during the period that the CorTemp® Disposable Temperature Sensor is within the body.
* Subjects hypomotility disorders of the gastrointestinal tract including but not limited to Ileus.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Cerebral Spinal Fluid (CSF) P-Tau measured with PET-MR | 4 Weeks
  CSF P-tau is associated with cortical tau uptake
18MK6240 binding amount measured with PET-MR | 2 weeks
  Tau binding in the brainstem is associated with increases in CSF OxA. PET-MR using 18MK6240 (PET Radiotracer for Imaging Neurofibrillary), which will be performed 1-4 weeks before the LP (visit 2).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Osorio, M.D, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Blessing EM, Parekh A, Betensky RA, Babb J, Saba N, Debure L, Varga AW, Ayappa I, Rapoport DM, Butler TA, de Leon MJ, Wisniewski T, Lopresti BJ, Osorio RS. Association between lower body temperature and increased tau pathology in cognitively normal older adults. Neurobiol Dis. 2022 Sep;171:105748. doi: 10.1016/j.nbd.2022.105748. Epub 2022 May 10. PMID 35550158